CLINICAL TRIAL: NCT01119404
Title: Hämeenlinna Metabolic Syndrome Research Program (HMS): Surrogate Indicators for Atherosclerosis in Men With Metabolic Syndrome, Coronary Heart Disease and Controls
Brief Title: Hämeenlinna Metabolic Syndrome Research Program: Surrogate Indicators for Atherosclerosis
Acronym: HMS-02
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanta-Häme Central Hospital (Other Government)
Collaborators: Linnan Klinikka Oy (Other); Mehiläinen Hämeenlinna, Finland (Unknown); Finnish Red Cross Blood Service (Other)
Responsible Party: Ari Palomäki, MD PhD, Central Hospital of Kanta-Häme
Other Study IDs: KHMetS-02-AP; HMS-02 (Other: Ethics Committee)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Metabolic Syndrome; Coronary Heart Disease
Keywords: Metabolic Syndrome; Coronary Heart Disease; Erectile Dysfunction; Arterial Elasticity; Oxidized Low Density Lipoprotein; Cardiovascular Diseases; Risk Assessment; Endothelial Dysfunction; Diabetes Mellitus; Surrogate Markers; Risk Factors
MeSH Terms: conditions — Metabolic Syndrome; Coronary Disease; Erectile Dysfunction; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, EDTA plasma, citrate plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Metabolic Syndrome: 120 men with metabolic syndrome
- Coronary Heart Disease (CHD): 120 men with angiographically verified CHD
- Control: 80 physically active men

SUMMARY:
Mechanisms that link metabolic syndrome to atherosclerosis are incompletely understood. As a part of Hämeenlinna Metabolic Syndrome Research Program (HMS) surrogate indicators for atherosclerosis are studied in 120 men with metabolic syndrome, 120 men with coronary heart disease and 80 physically active controls and in different settings.

DETAILED DESCRIPTION:
Accumulation of oxidized low-density lipoproteins (LDL) in the intimae of arteries together with risk factors known to enhance atherosclerosis, damage the endothelium of the arterial wall. Dysfunction of the endothelium leads into loss of elasticity of the artery. Surrogate indicators of atherosclerosis might be seen already in the early phase of otherwise subclinical arterial disease.

In this study, we investigate calculated risk of the subjects (SCORE, FINRISK, Framingham score), platelet function and surrogate indicators for atherosclerosis like erectile dysfunction, plasma levels of oxidized LDL, arterial elasticity and biochemical markers for endothelial damage and dysfunction in different settings (case-only and case-control).

ELIGIBILITY:
Inclusion Criteria:

Group 1: Metabolic syndrome

* 120 Finnish men with metabolic syndrome (MetS) defined according to National Cholesterol Education Program (NCEP) Adult Treatment Panel III
* MetS diagnosed in routine health examination and laboratory tests
* Age: 30 to 65 years

Group 2: Coronary heart disease (CHD)

* 120 Finnish men with angiographically proven CHD
* Age: 30 to 65 years

Group 3: Control

* 80 Finnish men
* Exercising physically more than three times a week and more than 30 minutes per exercise on regular basis
* Never been studied or treated because of cardiovascular disease
* Age: 30 to 65 years

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2003-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ari K Palomäki, MD PhD, Study Director — Central Hospital of Kanta-Häme; Kalevi Oksanen, MD PhD, Study Director — Central Hospital of Kanta-Häme
Locations (4):
- Finland (4):
  - Linnan Klinikka, Hämeenlinna
  - Mehiläinen Hämeenlinna, Hämeenlinna
  - Central Hospital of Kanta-Häme, Hämeenlinna
  - Finnish Red Cross Blood Transfusion Service, Helsinki

REFERENCES:
- [Derived] Saarinen HJ, Lahtela J, Mahonen P, Palomaki A; Hameenlinna Metabolic Syndrome Research Program Study Group. The association between inflammation, arterial stiffness, oxidized LDL and cardiovascular disease in Finnish men with metabolic syndrome - a 15-year follow-up study. BMC Cardiovasc Disord. 2024 Mar 15;24(1):162. doi: 10.1186/s12872-024-03818-x. PMID 38491429
- [Derived] Pohjantahti-Maaroos H, Palomaki A, Kankkunen P, Husgafvel S, Knuth T, Vesterinen K, Oksanen K. Arterial elasticity and oxidized LDL among men with metabolic syndrome and different 10-year cardiovascular risk estimated by FINRISK and SCORE models. Ann Med. 2012 Aug;44(5):503-12. doi: 10.3109/07853890.2011.590520. Epub 2011 Jul 4. PMID 21726125
- [Derived] Pohjantahti-Maaroos H, Palomaki A, Hartikainen J. Erectile dysfunction, physical activity and metabolic syndrome: differences in markers of atherosclerosis. BMC Cardiovasc Disord. 2011 Jun 27;11:36. doi: 10.1186/1471-2261-11-36. PMID 21707993